CLINICAL TRIAL: NCT00974441
Title: A Relative Bioavailability Study of 500 mg Divalproex Sodium Extended Release Tablets Under Fasting Conditions
Brief Title: Divalproex Sodium 500 mg Extended Release Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R06-0441
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Divalproex Sodium (Experimental): 500 mg Extended Release Tablet
  Interventions: Drug: Divalproex Sodium
- Depakote® (Active Comparator): 500 mg Extended Release Tablet
  Interventions: Drug: Depakote®

INTERVENTIONS:
Drug: Divalproex Sodium — 500 mg Extended Release Tablet
  Arms: Divalproex Sodium
Drug: Depakote® — 500 mg Extended Release Tablet
  Arms: Depakote®

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 500 mg Divalproex Sodium (equivalent to 500 mg Valproic Acid) Extended Release Tablets with that of Depakote® ER Tablets following a single oral dose (1 x 500 mg tablet) in healthy adult subjects administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria

* Subjects who have completed the screening process within 28 days prior to Period 1 dosing
* Subjects who are healthy adult men and women 18 years of age or older at the time of dosing.
* Subjects who have a body mass index (BMI) between 19-30 kg/m2, inclusive, and weigh at least 110 lbs.
* Subjects who are healthy as documented by the medical history, physical examination (including bur may not be limited to and evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems), vital sign assessments, 12-lead electrocardiogram (ECG), clinical laboratory assessments, and by general observations. Any abnormalities/deviations from the normal range that might be considered clinically relevant by the study physician and investigator will be evaluated for individual cases, documented in study files and agreed upon by both the study physician and investigator prior to enrolling the subject in this study and for continued enrollment.
* Female subjects of postmenopausal (no menses) status for at least 1 year and has a serum FSH level greater than or equal to 30 mIU/mL or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).

Exclusion Criteria

* Subjects who report receiving any investigational drug within 30 days prior to Period 1 dosing.
* Subjects who report any presence or history of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease as determined by the clinical investigator(s).
* Subjects whose clinical laboratory test values outside the accepted reference range and when confirmed on re-examination is deemed to be clinically significant.
* Subjects who demonstrate a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Subjects who report a history or allergic response(s) to divalproex or related drugs.
* Subjects who report the use of any systemic prescription medication in the 14 days prior to Period 1 dosing.
* Subjects who report the use of any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period 1 dosing.
* Subjects who report a history of clinically significant allergies including drug allergies.
* Subjects who report a clinically significant illness during the 4 weeks prior to Period 1 dosing (as determined by the clinical investigators).
* Subjects who report a history of drug or alcohol addiction or abuse within the past year.
* Subjects who demonstrate a positive drug abuse screen for this study prior to Period 1 administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Cmax - Maximum Observed Concentration | Blood samples collected over 72 hour period
AUC0-inf - Area under the concentration-time curve from time zero to infinity (extrapolated) | Blood samples collected over 72 hour period
AUC0-t - Area under the concentration-time curve from time zero to time of last quantifiable concentration (per participant) | Blood samples collected over 72 hour period

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States